CLINICAL TRIAL: NCT05152303
Title: Efficacy and Safety of Remimazolam Tosilate for Injection for Sedation in the Intensive Care Unit (ICU) - a Multicenter, Randomized, Single Blind, Dose Finding Phase II Clinical Trial
Brief Title: A Study of Remimazolam Tosilate for Sedation in the ICU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR7056-205
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Sedation in the ICU

STUDY DESIGN:
Intervention Model Description: This is a Multicenter, Randomized, Single Blind, Dose Finding, Phase II Clinical Trial to explore the optimal dose regimen of Remimazolam Tosilate for Injection for sedation in the ICU, as well as preliminarily evaluate the efficacy and safety of Remimazolam Tosilate for Injection for sedation in the ICU
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A：Remimazolam Tosilate (Experimental)
  Interventions: Drug: Remimazolam Tosilate
- B：Remimazolam Tosilate (Experimental)
  Interventions: Drug: Remimazolam Tosilate

INTERVENTIONS:
Drug: Remimazolam Tosilate — Loading dose: 0.08mg/kg IV of Remimazolam Tosilate, Maintenance dose: IV remimazolam tosilate, dose range 0-2.0mg/kg/h, increment or decrement of 0.1mg/kg/h
  Arms: A：Remimazolam Tosilate
Drug: Remimazolam Tosilate — Loading dose: 0.08mg/kg, Drug: Propofol Injection Maintenance dose: IV remimazolam tosilate, dose range 0-2.0mg/kg/h, increment or decrement of 0.2mg/kg/h IV of Propofol Injection
  Arms: B：Remimazolam Tosilate

SUMMARY:
The purpose of this study is to explore the optimal dose regimen of Remimazolam Tosilate for Injection for sedation in the ICU, as well as preliminarily evaluate the efficacy and safety of Remimazolam Tosilate for Injection for sedation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their guardians are able to provide a written informed consent
2. Subjects have been treated with endotracheal intubation and mechanical ventilation, and is expected to receive sedation after randomization. The target level and duration of sedation meet the criteria
3. Meet the age criteria, male or female
4. Meet the BMI criteria

Exclusion Criteria:

1. Deep sedation is required, or continuous sedation is not needed during the study process
2. Subjects with a history of severe cardiovascular disease, or cerebrovascular disease, or neurological disease, or mental illness
3. Subjects with a history of drug abuse
4. Subjects after neurosurgery operation
5. Organ failure before randomization
6. Abnormal values of the laboratory examination
7. Abnormal blood pressure and heart rate during screening
8. Allergic to relevant drugs ingredient or component
9. Pregnant or nursing women
10. Subjects who has participated in clinical trials of other interventions recently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Rate of sedation success, sedation success is defined as the percentage of time maintaining target sedation in the entire drug administering time ≥ 70% without rescue sedation | within 24 hours after administration of research drug

SECONDARY OUTCOMES:
Percentage of time maintaining target sedation in the entire drug administering time. | within 24 hours after administration of research drug
Percentage of subjects receiving rescue sedation and the average dosage of rescue sedation | within 24 hours after administration of research drug
Percentage of subjects receiving rescue analgesia and the average dosage of rescue analgesiaassessment time point after drug administering. | within 24 hours after administration of research drug
The number of times to change the infusion rate | within 24 hours after administration of research drug
Wake-up time. | within 8 hours after stopping the research drug
Evaluation of nursing difficulty. | follow-up period (approx. 5-10 minutes)
Mechanical ventilation time. | at the time of extubation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu N, Jiang Z, Nie Y, Zuo L, Chen C, Si X, Liu Q, Chen M, Guan X. Study Protocol of a Multicenter, Randomized, Single-Blind Trial: Efficacy and Safety of Remimazolam Tosylate for Sedation in ICU Patients. Adv Ther. 2023 May;40(5):2524-2533. doi: 10.1007/s12325-023-02456-7. Epub 2023 Mar 15. PMID 36920745